CLINICAL TRIAL: NCT01289639
Title: Insulin Resistance in Non-alcoholic Fatty Liver Disease (Protocol Drug Change From Project Career Development Award (CDA)-2-044-08S)
Brief Title: Insulin Resistance in Non-alcoholic Fatty Liver Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment in intervention study. Baseline data published.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CDA-2-044-08S-2
Record Dates: First submitted 2011-01-21; First posted 2011-02-04 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Fatty Liver
Keywords: non-alcoholic fatty liver disease; non-alcoholic steatohepatitis; insulin resistance; pioglitazone; fenofibrate
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — Fenofibrate; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): matching placebo 1 po qd
  Interventions: Drug: placebo
- Fenofibrate (Experimental): micronized fenofibrate 200 mg 1 po qd
  Interventions: Drug: fenofibrate
- Pioglitazone (Experimental): pioglitazone 30 mg po qd
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: fenofibrate — micronized fenofibrate 200 mg 1 po qd
  Other Names: micronized fenofibrate
  Arms: Fenofibrate
Drug: pioglitazone — pioglitazone 30 mg po qd
  Other Names: Actos
  Arms: Pioglitazone
Drug: placebo — placebo 1 capsule po qd
  Arms: Placebo

SUMMARY:
The study is designed to investigate the relationship between insulin resistance and non-alcoholic fatty liver disease (NAFLD) and to investigate potential mechanisms underlying insulin resistance in NAFLD by determining associations between hepatic and peripheral insulin sensitivity, hepatic steatosis, dyslipidemia, inflammatory cytokines, glucose metabolism, beta-cell function and body fat distribution.

DETAILED DESCRIPTION:
NAFLD and nonalcoholic steatohepatitis (NASH) are common liver disorders that are strongly associated with obesity, type 2 diabetes and dyslipidemia. The underlying pathophysiology of fatty infiltration of the liver is thought to be related to insulin resistance, which is an almost universal finding in patients with NAFLD. It is also possible that fat infiltration and inflammation in the liver may impair insulin sensitivity, either locally in the liver, or peripherally via the actions of inflammatory cytokines. We hypothesize that insulin resistance is a major causal factor leading to fat deposition in the liver and NAFLD, and thus interventions aimed at improving insulin sensitivity will result in a reduction of hepatic inflammation and steatosis.

Specific Aim 1: To determine in a cross-sectional study whether NAFLD is associated with altered peripheral and hepatic insulin sensitivity and to study their relationships with hepatic steatosis, dyslipidemia, inflammatory cytokines, glucose metabolism, beta-cell function and body fat distribution. Specific Aim 2: To determine in a 6 month placebo-controlled double-blinded treatment study if treatment with pioglitazone, an insulin sensitizer, or fenofibrate, a triglyceride lowering agent, will improve both hepatic as well as peripheral insulin sensitivity and thereby improve hepatic steatosis and inflammation in subjects with NAFLD.

The results of the proposed study will have important implications for our understanding of the mechanisms underlying insulin resistance and abnormalities in lipid and glucose metabolism in subjects with NAFLD and for the design of future studies aimed at the prevention and treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

Control subjects: nl liver enzymes and no history of liver disease Case subjects: NAFLD on liver biopsy within the past 3 years or presumed NAFLD with otherwise unexplained elevated alanine aminotransferase (ALT) and fatty liver by computerized tomography (CT) scan or ultrasound

* Able to comply with taking 1 pill a day for 6 months and follow-up safety visits

Exclusion Criteria:

* Cases: cirrhosis on liver biopsy or by clinical exam or fibrosis score
* Causes of liver dysfunction other than NASH
* Use of medications associated with hepatic steatosis:

  * glucocorticoids
  * estrogens
  * tamoxifen
  * amiodarone
  * accutane
  * sertraline
* Use of medications that cause insulin resistance:

  * niacin
  * glucocorticoids
  * anti-HIV drugs or atypical antipsychotics
* Use of lipid-lowering medications except stable dose statin
* Use of anti-NASH drugs such as ursodeoxycholic acid, betaine milk thistle
* Use of coumadin
* Use of nitrates
* Significant alcohol consumption: Average >20 grams/day
* In subjects with diabetes, a hemoglobin A1c (HbA1c) >7.5% or use of insulin, metformin, rosiglitazone or pioglitazone
* Liver transaminases: ALT >5x upper limit of normal,
* Iron saturation >50%
* Creatinine >1.5 mg/dl for men and >1.4 mg/dl for women
* Hematocrit <33%
* Pregnancy or lactation
* Significant weight loss within the past 6 months or since the liver biopsy
* History of significant coronary artery disease or congestive heart failure, retinopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-10; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Utzschneider, MD, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States

REFERENCES:
- [Result] Utzschneider KM, Largajolli A, Bertoldo A, Marcovina S, Nelson JE, Yeh MM, Kowdley KV, Kahn SE. Serum ferritin is associated with non-alcoholic fatty liver disease and decreased Beta-cell function in non-diabetic men and women. J Diabetes Complications. 2014 Mar-Apr;28(2):177-84. doi: 10.1016/j.jdiacomp.2013.11.007. Epub 2013 Nov 26. PMID 24360972
- [Result] Kratz M, Marcovina S, Nelson JE, Yeh MM, Kowdley KV, Callahan HS, Song X, Di C, Utzschneider KM. Dairy fat intake is associated with glucose tolerance, hepatic and systemic insulin sensitivity, and liver fat but not beta-cell function in humans. Am J Clin Nutr. 2014 Jun;99(6):1385-96. doi: 10.3945/ajcn.113.075457. Epub 2014 Apr 16. PMID 24740208

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: matching placebo for fenofibrate 1 capsule po qd
  matching placebo for pioglitazone 1 capsule po qd
- Arm 2: micronized fenofibrate 200 mg 1 po qd
  matching placebo for pioglitazone 1 po qd
- Arm 3: pioglitazone 30 mg po qd
  matching placebo for fenofibrate 1 po qd
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 5 | 6 | 0
Completed | 4 | 6 | 0
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects recruited with known NAFLD or NASH.
Groups:
- Arm 1: matching placebo for fenofibrate 1 po qd
  matching placebo for pioglitazone 1 po qd
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 5 | 6 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (7.3) | 54.17 (5.08) |  | 51.91 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 |  | 4
  Male | 3 | 4 |  | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Liver/Spleen Ratio Measured as the Ratio in Hounsfield Units Between the Liver and the Spleen on Computed Tomography (CT) Scan
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 6 | 0
ratio | .85 (.08) | .60 (.17) |

2. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Levels
Time Frame: 0-6 months
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 6 | 0
U/L | -11.5 (12.9) | -15.2 (4.5) |

3. Secondary Outcome: Change in Liver/Spleen Ratio Measure by the Density Ratio in Hounsfield Units Between the Liver and the Spleen by CT
Time Frame: 0-6 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 6 | 0
ratio | .09 (.10) | -0.16 (0.1) |

4. Secondary Outcome: Change in Peripheral Insulin Sensitivity
Description: Change in the rate of glucose disposal (Rd) during the low dose clamp. During a clamp procedure, insulin is infused at a dose based on body size and a glucose solution is infused and the rate adjusted every 5 minutes based on a blood glucose reading to maintain the blood glucose stable at 90 mg/dl (normal level). Using glucose isotopes and the rate of the glucose infusion, we are then able to calculate how much glucose the liver is producing and how much glucose is being taken up into tissues. This provides a measure of insulin sensitivity.
Time Frame: 0-6 months
Measure: Mean (Standard Error); unit: mg/minute/kg lean mass
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 5 | 0
mg/minute/kg lean mass | 0.21 (0.51) | -0.42 (0.49) |

5. Secondary Outcome: Change in Intra-abdominal Fat Area by CT Scan
Time Frame: 0-6 months
Measure: Mean (Standard Error); unit: mm2
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 6 | 0
mm2 | 885 (874) | 108 (3416) |

6. Secondary Outcome: Change in Hepatic Insulin Sensitivity
Description: Hepatic insulin sensitivity was determined using stable glucose isotope measurements during the low dose hyperinsulinemic euglycemic clamp to determine the rate of endogenous glucose production in the fasting state and in response to a low dose glucose infusion. The ability of insulin to suppress glucose, which is mainly produced by the liver, thus provides a measure of hepatic insulin sensitivity and is expressed as a percentage of the basal state. Change in the ability of low dose insulin to suppress endogenous glucose production during a labeled hyperinsulinemic euglycemic clamp.
Time Frame: 0-6 months
Measure: Mean (Standard Error); unit: % change from baseline
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 5 | 0
% change from baseline | 23.3 (7.8) | 4.9 (9.3) |

ADVERSE EVENTS:
Time Frame: Baseline and monthly.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 3/5 | 4/6 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=5) | Arm 2 (N=6) | Arm 3 (N=0)
leg edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
vasovagal reaction (General disorders) | 2 (2) | 0 (0) | 0 (0)
gout attack (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
increased serum creatinine (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to low enrollment, the study was stopped prematurely. Due to the low number of subjects enrolled, statistical analysis was not possible on the intervention study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No